CLINICAL TRIAL: NCT03301909
Title: Development of Applications of PillCam™ Endoscopy and Patency Systems and Clinical Evaluation of Their Performance in Healthy Volunteers ("HEIGHT" Study)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study purposes and objectives have shifted
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MDT16024
Record Dates: First submitted 2017-09-29; First posted 2017-10-04 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PillCam™ Endoscopy System (Experimental): PillCam™ Endoscopy System consists of the following subunits:
  * PillCam™ Capsule products' family:
    1. PillCam™ COLON 2
    2. PillCam™ UGI (upper gastrointestinal)
    3. PillCam™ SB3 (small bowel 3)
    4. PillCam™ Crohn's capsule
  * Patency capsule: PillCam™ Patency capsule
  All the bellow system subunits are part of the Pillcam™ systems:
  * PillCam™ Recorder
  * PillCam™ Sensor Arrays & Sensor Belt
  * PillCam™ Software v. 9
  * Workstation unit
  Interventions: Device: PillCam™ Endoscopy System; Drug: Bowel prep combination

INTERVENTIONS:
Device: PillCam™ Endoscopy System — Subject may be assigned to any procedure involving modification of any of the PillCam™ Endoscopy System component as listed in the arm description.
Drug: Bowel prep combination — Subject may be assigned to any bowel preparation combination.

SUMMARY:
This is a feasibility, prospective, single center, open label, uncontrolled clinical study, to evaluate the safety and preliminary efficacy of the different R&D changes made and implemented in the existing PillCam Capsule products family, PillCam Endoscopy System subunits, the Patency system and bowel preparation procedure.

DETAILED DESCRIPTION:
The study consists of a screening - enrollment phase, a possible preparation phase followed by the PillCam Endoscopy or Patency procedure visit and a post procedure telephone, follow up visit.

Subjects may be assigned to any of the sub-assays done within this study as long as they fulfill all the inclusion and exclusion criteria and depends on their availability and their willingness to participate in a specific sub-assay.

Each subject may participate in up to 15 sub-assays during his/her participation in the study, each ingestion will be separated in between by at least two weeks interval. A following capsule may be ingested only upon verification of previous capsule excretion. Subjects can participate in a specific sub-assay only once.

In general, under the study protocol, per a single procedure, each subject will undergo a possible preparation phase followed by the PillCam endoscopy or Patency procedure and telephone follow up visit. Overall the expected duration for subject's participation in the study is expected to be up to 10 years, until subject will complete participation in up to 15 sub-assays.

Subject may withdraw consent at any time and will be considered as completed once completed at least one capsule ingestion (PillCam or Patency) or completed one of the possible procedures which are not involving capsule ingestion during the study period.

ELIGIBILITY:
Inclusion Criteria:

1. Subject either male or female is 45-85 years of age.
2. The subject is in good general health to enable participation in the study.
3. The subject received an explanation and understands the nature of the study and agrees to provide written informed consent.

Exclusion Criteria:

1. Subject has dysphagia or any swallowing disorder.
2. Subject is known or is suspected to suffer from intestinal obstruction or stricture (symptoms such as severe abdominal pain with accompanying nausea or vomiting).
3. Subject with known gastrointestinal motility disorders.
4. Subjects with known or suspected delayed gastric emptying.
5. Subject has known or suspected Crohn's disease, other inflammatory bowel disease, perforations or structural disorders of the gut wall.
6. Subject has diabetes.
7. Subject has undergone certain prior abdominal surgery of the gastrointestinal tract, (other than uncomplicated appendectomy or uncomplicated cholecystectomy) which may interfere with the study, such as small bowel or colonic resection. This will be evaluated by the investigator.
8. Subject has any allergy or other contraindication to any materials including preparation used prior, during or after capsule endoscopy in the study.
9. Subject is expected to undergo MRI examination within 7 days after ingestion of the capsule.
10. Subject has severe congestive heart failure or known renal or hepatic insufficiency.
11. Subject has a cardiac pacemakers or other implanted electromedical devices.
12. Subject has any condition, which according to the investigators judgment, precludes compliance with study and/or device instructions.
13. Females who are pregnant or nursing at the time of screening and/or during the study period, or are of child bearing potential without medically acceptable methods of contraception.
14. Subject is currently participating in another clinical study that may directly or indirectly affect the results of this study.
15. Subject is considered to be part of a vulnerable population (e.g. prisoners or those without sufficient mental capacity).

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 694 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2023-03-27 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
All device related Adverse events will be collected and reported in order to assess the device safety. | Up to 10 years
  All device related Adverse events will be reported by number, type, seriousness, severity and duration. All device related adverse events will be captured, regardless of severity.

SECONDARY OUTCOMES:
Assessment of raw data generation in the data recorder by confirming presence of the procedure raw data output files (technical outcome) | Up to 10 years
  A PillCam procedure will be assessed for raw data generation in the data recorder (similar to standard of care procedure), by confirming presence of the procedure output files (technical outcome). A nominal scale of Yes/No will be used to determine whether the raw data has been generated by the data recorder or not.

CONTACTS AND LOCATIONS:
Overall Officials: Wisam Sbeit, M.D, Principal Investigator — Galil MC, Nahariya
Locations (1):
- Medtronic - Glilee Medical Center, Yokneam Illit, Israel

IPD SHARING:
Plan to Share IPD: No